CLINICAL TRIAL: NCT02462746
Title: The Effect of Cysteine, Tryptophan and Tyrosine Supplements on Breast Milk
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Jeff Meyer, Canada Research Chair, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100-2014
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: Postpartum; Dietary Supplements; Breastfeeding Women
MeSH Terms: interventions — Cysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No supplement (No Intervention): This group subjects will not receive the supplement
- 1.5 gram of l-cysteine (Active Comparator): Intervention: single dose of 1.5 g L-Cysteine.
  Interventions: Dietary Supplement: L-Cysteine
- 3 grams of l-cysteine (Active Comparator): Intervention: single dose of 3.0 g L-Cysteine.
  Interventions: Dietary Supplement: L-Cysteine

INTERVENTIONS:
Dietary Supplement: L-Cysteine — The trade name is New Root Herbal Inc.
  Other Names: Cysteine
  Arms: 1.5 gram of l-cysteine; 3 grams of l-cysteine

SUMMARY:
The purpose of this project is to study the effect of dietary supplementation with a natural health product (NHP) with a focus on its effects on its levels in breast milk.

DETAILED DESCRIPTION:
The effect of oral cysteine on its levels in breast milk and plasma will be measured in breast feeding mothers.

The investigators will not be studying tryptophan and tyrosine in this study. The title is an overview title left over from other past studies (but the investigators are only assessing cysteine at this time).

ELIGIBILITY:
Inclusion Criteria:

* Subjects would be healthy mothers who are breastfeeding at the moment, but plan to stop at the time of study
* The subject, as reported, should be in a good health
* The subject is not taking any medication
* The subject is not taking any investigational medicinal product within 8 weeks prior to dosing
* The subject does not have any known hypersensitivity to components in the proposed treatment
* The subject does not have a history of severe drug allergy or drug hypersensitivity

Other general medical requirements for inclusion:

* Age 18 to 45
* BMI 19 to 40 (kg/m2)
* Resting pulse between 45 and 100 bpm
* Systolic blood pressure between 91 and 139 mmHg (inclusive)
* Diastolic blood pressure between 51 and 90 mmHg (inclusive)
* Orthostatic blood pressure change <20 mmHg (based on the difference between supine and standing (1 minute) systolic blood pressure)
* The subject is in good health based on their report and answer to general health questionnaire

Exclusion Criteria:

* The subject has taken any investigational medicinal product within 8 weeks prior to dosing
* The subject is pregnant (based upon urine pregnancy test at time of screening and day of supplement intake)
* The subject has known hypersensitivity to components in the proposed treatment or to related compounds
* The subject has a history of severe drug allergy or drug hypersensitivity involving an anaphylactic reaction i.e. shortness of breath and/or reduced blood pressure
* Subjects who are smoking more than one package of cigarette per day will be excluded from the study
* The subject decides to breastfeed the infant on the study day

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Breast milk cysteine levels | The main protocol occurs of 10 hours of time when the pharmacokinetics of the amino acid are measured.
  measurement of amino acid before and after acute administration over a 10 hour period
  * The first visit would be the screening visit, which the subjects will be evaluated for general health status through a standardized health questionnaire. A urine test will be done in order to screen for any drug use.
  * On the second visit, each subject would be tested for plasma levels of the amino acid during the day. In addition breast milk will be tested in order to examine the effect of these supplements on the amino acid contents of the breast milk at few time points on both days.

SECONDARY OUTCOMES:
plasma cysteine levels | These are sampled over 10 hours before and after administration of cysteine
  These are the acute changes in plasma cysteine levels over 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Meyer, MD,PhD, Principal Investigator — Centre for Addiction and Mental Health, Research Imaging Centre, Toronto, Ontario, Canada M5T 1R8
Locations (1):
- Research Imaging Centre, Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://camh.ca/research